CLINICAL TRIAL: NCT00020462
Title: Active Specific Immunotherapy for Follicular Lymphomas With Liposomes Containing Tumor-Derived Antigen and IL-2
Brief Title: Vaccine Therapy Plus Interleukin-2 in Treating Patients With Stage III, Stage IV, or Recurrent Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068505; NCI-01-C-0069; NCT00008996 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-08-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2008-12

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — aldesleukin; FANG vaccine

INTERVENTIONS:
Biological: aldesleukin
Biological: autologous tumor cell vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to kill tumor cells. Combining vaccine therapy with interleukin-2 may be a more effective treatment for follicular lymphoma .

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy plus interleukin-2 in treating patients who have stage III, stage IV, or recurrent follicular lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety of immunotherapy with autologous tumor cell vaccine and interleukin-2 in patients with stage III, IV, or recurrent follicular lymphoma.
* Determine the clinical response of patients treated with this regimen.
* Assess the immune response of patients treated with this vaccine.

OUTLINE: This is a multicenter study. Patients are stratified according to prior therapy (no prior biologic therapy or chemotherapy for lymphoma vs prior prednisone, doxorubicin, cyclophosphamide, and etoposide (PACE) chemotherapy). Patients without prior therapy are further stratified according to accessibility of lymph nodes (easily accessible (stratum Ia) vs not easily accessible (stratum Ib)).

All patients undergo lymph node biopsy to obtain tissue for vaccine manufacture. Treatment begins approximately 1 month after biopsy.

* Stratum Ia: Patients receive autologous tumor cell vaccine and interleukin-2 (IL-2) intranodally and subcutaneously (SC) on day 1.
* Stratum Ib and stratum II: Patients receive autologous tumor cell vaccine and IL-2 SC on day 1.

Treatment in each stratum continues every 4 weeks for a maximum of 5 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 and 4 months, every 3 months for 1 year, and every 6 months thereafter until relapse or progression of disease.

PROJECTED ACCRUAL: A total of 20 patients (10 per stratum) will be accrued for this study within 1.5-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven follicular center cell lymphoma with surface immunoglobulin (Ig) M, G, or A phenotype

  * Grade I (follicular small cleaved cell)
  * Grade II (follicular mixed small and large cell)
  * Grade III (follicular large cell)
* Stage III, IV, or recurrent disease
* Previously untreated with chemotherapy or monoclonal antibody therapy OR
* Recurrent, residual disease or progressive disease after prior prednisone, doxorubicin, cyclophosphamide, and etoposide (PACE) chemotherapy
* Peripheral lymph node of at least 2 cm and accessible for biopsy/harvest
* No primary or secondary CNS lymphoma
* Must not have any of the following:

  * Rapidly progressing lymphadenopathy
  * Bone marrow failure secondary to lymphoma
  * B symptoms
  * Neurovascular or organ compromise secondary to lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 1 year

Hematopoietic:

* Not specified

Hepatic:

* ALT/AST no greater than 3.5 times upper limit of normal
* Bilirubin no greater than 1.5 mg/dL unless secondary to Gilbert's disease
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* HIV negative
* No active infection
* No other prior or concurrent malignancy except curatively treated squamous cell or basal cell skin cancer or effectively treated carcinoma in situ of the cervix
* No medical or psychiatric condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No other concurrent biologic therapy for lymphoma

Chemotherapy:

* See Disease Characteristics
* At least 3 months since prior PACE chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 2 weeks since prior steroid treatment
* Less than 2 months of prior prednisone
* No concurrent endocrine therapy for lymphoma

Radiotherapy:

* Prior radiotherapy to no more than 1 site allowed
* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Lymph node biopsy performed within past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Sattva S. Neelapu, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States

REFERENCES:
- [Result] Neelapu SS, Gause BL, Harvey L, Lee ST, Frye AR, Horton J, Robb RJ, Popescu MC, Kwak LW. A novel proteoliposomal vaccine induces antitumor immunity against follicular lymphoma. Blood. 2007 Jun 15;109(12):5160-3. doi: 10.1182/blood-2006-12-063594. Epub 2007 Mar 5. PMID 17339422